CLINICAL TRIAL: NCT01983774
Title: Effect of Proton Pump Inhibitors on CF Exacerbations
Brief Title: Effect of Proton Pump Inhibitors on CF Pulmonary Exacerbations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Emily DiMango, MD, Associate Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAC5640
Record Dates: First submitted 2013-11-06; First posted 2013-11-14 (Estimated); Results first posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-01

CONDITIONS: Cystic Fibrosis
Keywords: CF
MeSH Terms: conditions — Cystic Fibrosis | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): A matching placebo (sugar pill) to esomeprazole 40mg twice daily
  Interventions: Drug: Placebo
- Esomeprazole (Active Comparator): Esomeprazole 40mg twice daily
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole
  Other Names: Nexium
  Arms: Esomeprazole
Drug: Placebo — Sugar pill
  Arms: Placebo

SUMMARY:
Gastroesophageal reflux disease (GERD) is a common problem in cystic fibrosis (CF). It may lead to worsening lung function and more respiratory infections for a person with CF. This study will look at treating GERD with a medication, esomeprazole. The medication stops stomach acid from being made. The study will see if there are fewer respiratory infections and improved lung function in patients with CF when taking esomeprazole.

DETAILED DESCRIPTION:
This is a randomized, placebo controlled intervention study in patients with CF who have a history of frequent exacerbations. Treatment duration is 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Cystic fibrosis
2. Age > 18 years
3. Stable maintenance medical regimen during the previous 6 weeks.
4. Negative pregnancy test (women of childbearing potential) at both screening and baseline visits.
5. Women of childbearing potential must be using medically acceptable contraception.
6. At least two respiratory exacerbations per year requiring oral and/or intravenous antibiotics for each of the two years prior to study entry, but no more than 4 exacerbations requiring intravenous antibiotics during either of those years.

Exclusion Criteria:

1. Previous anti-reflux or peptic ulcer surgery,
2. Use of proton pump inhibitor (PPI) within the past two weeks
3. Pulmonary exacerbation requiring antibiotics within the previous 2 weeks
4. Parenteral hyperalimentation
5. Cigarette smoking
6. Treatment with azoles, iron, anti-coagulants, digitalis
7. Use of any investigative drugs within the previous month.
8. Use of over the counter acid suppressor agents (not including acid neutralizers)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily DiMango, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Cystic Fibrosis Center, New York, New York, United States

REFERENCES:
- [Derived] Ng SM, Moore HS. Drug therapies for reducing gastric acidity in people with cystic fibrosis. Cochrane Database Syst Rev. 2021 Apr 27;4(4):CD003424. doi: 10.1002/14651858.CD003424.pub5. PMID 33905540
- [Derived] Hurley MN, Smith S, Forrester DL, Smyth AR. Antibiotic adjuvant therapy for pulmonary infection in cystic fibrosis. Cochrane Database Syst Rev. 2020 Jul 16;7(7):CD008037. doi: 10.1002/14651858.CD008037.pub4. PMID 32671834
- [Derived] Dimango E, Walker P, Keating C, Berdella M, Robinson N, Langfelder-Schwind E, Levy D, Liu X. Effect of esomeprazole versus placebo on pulmonary exacerbations in cystic fibrosis. BMC Pulm Med. 2014 Feb 15;14:21. doi: 10.1186/1471-2466-14-21. PMID 24528942
- See also: Results Reference — https://bmcpulmmed.biomedcentral.com/articles/10.1186/1471-2466-14-21

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-one participants were assessed for eligibility. Of those, four were excluded (two did not meet inclusion criteria and two declined participation). Seventeen participants were randomized.
Groups:
- Esomeprazole: Esomeprazole 40mg twice daily
  Esomeprazole
Period: Overall Study
Arm/Group | Esomeprazole | Placebo
Started | 9 | 8
Completed | 8 | 7
Not Completed | 1 | 1
Not completed — Lung Transplant | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Esomeprazole: Esomeprazole 40 mg twice daily
- Placebo: A matching placebo (sugar pill) to esomeprazole 40 mg twice daily.
- Total: Total of all reporting groups
Arm/Group | Esomeprazole | Placebo | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.72 (9.6) | 32.81 (5.84) | NA (NA) — Total mean age (and standard deviation) were not calculated upon initial data analysis. The data set was destroyed and no longer exists. The data are not available and therefore totals cannot be calculated.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 8 | 17
FEV1 [Mean (Standard Deviation); unit: percent predicted] | 58 (19) | 46 (21) | NA (NA) — Total mean FEV1 (and standard deviation) were not calculated upon initial data analysis. The data set was destroyed and no longer exists. The data are not available and therefore totals cannot be calculated.
Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: Percent Predicted] | 74 (20) | 71 (16) | NA (NA) — Total mean FVC (and standard deviation) were not calculated upon initial data analysis. The data set was destroyed and no longer exists. The data are not available and therefore totals cannot be calculated.
Number of exacerbations in the past two years [Mean (Standard Deviation); unit: Count of exacerbations] | 4 (0) | 5.5 (1.4) | NA (NA) — Total mean number of exacerbations (and standard deviation) were not calculated upon initial data analysis. The data set was destroyed and no longer exists. The data are not available and therefore totals cannot be calculated.

OUTCOME MEASURES:

1. Primary Outcome: Time to First Pulmonary Exacerbation
Description: Time to need for oral or intravenous antibiotics for treatment of a pulmonary exacerbation is the primary outcome measure.
Time Frame: 36 weeks
Population: Values per arm for time to first pulmonary exacerbation cannot be reported. The data set was destroyed and no longer exists. The only available results exist as a figure within the study publication.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 9 | 8
Weeks | NA (NA) — Time to first pulmonary exacerbation for esomeprazole arm cannot be reported. The data set was destroyed and no longer exists. The only available results exist as a figure within the study publication. | NA (NA) — Time to first pulmonary exacerbation for placebo arm cannot be reported. The data set was destroyed and no longer exists. The only available results exist as a figure within the study publication.

2. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1)
Description: Forced Expiratory Volume in one second (FEV1) as measured by spirometry
Time Frame: 36 weeks
Population: Values per arm for FEV1 cannot be reported. The data set was destroyed and no longer exists. The only available results exist as a figure within the study publication.
Measure: Mean (Standard Deviation); unit: percentage of predicted
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 9 | 8
percentage of predicted | NA (NA) — Values for the esomeprazole arm cannot be reported. The data set was destroyed and no longer exists. The only available results exist as a figure within the study publication. | NA (NA) — Values for the placebo arm cannot be reported. The data set was destroyed and no longer exists. The only available results exist as a figure within the study publication.

3. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Forced Vital Capacity percent predicted
Time Frame: 36 weeks
Population: Values per arm for FVC cannot be reported. The data set was destroyed and no longer exists. The only available results exist as a figure within the study publication.
Measure: Mean (Standard Deviation); unit: percentage of predicted
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 9 | 8
percentage of predicted | NA (NA) — Values for the esomeprazole arm cannot be reported. The data set was destroyed and no longer exists. The only available results exist as a figure within the study publication. | NA (NA) — Values for the placebo arm cannot be reported. The data set was destroyed and no longer exists. The only available results exist as a figure within the study publication.

4. Secondary Outcome: Number of Exacerbations
Description: Exacerbation defined as initiation of treatment with intravenous or oral antibiotics for 7 or more days based on respiratory symptoms
Time Frame: 36 weeks
Population: Values per arm for number of exacerbations cannot be reported. The data set was destroyed and no longer exists. The only available results exist in the study publication.
Measure: Mean (Standard Deviation); unit: Number of exacerbations
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 9 | 8
Number of exacerbations | NA (NA) — Values for the esomeprazole arm cannot be reported. The data set was destroyed and no longer exists. The only available results exist as listed in the study publication. | NA (NA) — Values for the placebo arm cannot be reported. The data set was destroyed and no longer exists. The only available results exist as listed in the study publication.

ADVERSE EVENTS:
Arm/Group | Esomeprazole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8

LIMITATIONS AND CAVEATS:
Study findings are limited by small sample size without adequate power to detect significant differences between participants treated with esomeprazole compared with placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes